CLINICAL TRIAL: NCT06475014
Title: Application of Knee Measurements on 3D Computed Tomography in Total Knee Replacement
Brief Title: Application of Knee Measurements on 3D CT in TKR
Status: Completed | Type: Observational
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Principal Investigator, Vo Sy Quyen Nang, MD, Vinmec Healthcare System
Other Study IDs: VOSCknee3D
Record Dates: First submitted 2024-06-13; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Knee Osteoarthritis; Knee Disease
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 365 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee with OA: Underwent Total Knee replacement Surgery, using 3D printed PSI,
  Interventions: Procedure: Total knee replacement

INTERVENTIONS:
Procedure: Total knee replacement — Mechanical Alignment Using PSI Pre and post-operative CT Scan

SUMMARY:
A 3D Computed Tomographic Study of Vietnamese Knee Morphology for Total knee Replacement

DETAILED DESCRIPTION:
There were controversies and inconsistent results regarding the effectiveness of PSI.

However, most authors used PSI from commercial manufacturers. From our view, the surgeon's involvement in PSI planning and design can affect the PSI's accuracy. Some other benefits of in-hospital PSI included the use of any type of implant without depending on the manufacturer's software system, faster and cheaper. Therefore, we conducted this study to evaluate the effect of in-hospital PSI in which the surgeons take part in the manufacturing job.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of knee osteoarthritis, grade III, IV
* Underwent total knee replacement using patient-specific intrumentation
* With pre and post-operative whole limb CT-Scanners

Exclusion Criteria:

* Paticipants with valgus knee deformity,
* A history of hip arthroplasty,
* Large bone defect that required augments.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with severe osteoarthritis of the knee who underwent primary TKA
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Radiology outcome | 30/06/2023
  Position of implants compare to the plan on CT, measure the discrepancies by degree
Clinical outcome, self-administered questionnaire | 30/06/2024
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) score, from 0-96, lower is better
Clinical outcome, by surgeon's evaluating | 30/06/2024
  The 2011 Knee Society Scoring System, from 0 to 100, higher is better

OTHER OUTCOMES:
AP-ML dimesion | 30/06/2023
  Size of knee on stimulated bone resection slice, AP and ML dimension in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Duong Dinh Toan, Ph.D, Study Chair — Hanoi Medical University
Locations (1):
- Vinmec Times City Hospital, Hanoi, Hai Ba Trung, Vietnam

IPD SHARING:
Plan to Share IPD: No